CLINICAL TRIAL: NCT04761952
Title: N-3 Polyunsaturated Fatty Acids Prevent Postoperative Recurrence of Crohn's Disease：a Prospective Randomized Controlled Trial
Brief Title: N-3 Polyunsaturated Fatty Acids Prevent Postoperative Recurrence of Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020ZSLYEC-292
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Polyunsaturated Acid Lipidosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Neuronal Ceroid-Lipofuscinoses | interventions — Azathioprine; Infliximab; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3PUFA treatment group (Experimental): On the basis of routine treatment, oral supplement of n-3PUFA was given to CD patients since 2-week-postoperative till 1-year-postoperative.
  Interventions: Drug: azathioprine; Drug: infliximab; Drug: N-3 Polyunsaturated Fatty Acids
- Conventional treatment group (Placebo Comparator): Treatment of azathioprine (daily orally) or infliximab (intravenously, at 0, 2,6 weeks with every 8-week-interval later) was given since 2-week-postoperative till 1-year-postoperative.
  Interventions: Drug: azathioprine; Drug: infliximab

INTERVENTIONS:
Drug: azathioprine — daily orally
  Other Names: AZA
Drug: infliximab — intravenously, at 0, 2,6 weeks with every 8-week-interval later
  Other Names: IFX
Drug: N-3 Polyunsaturated Fatty Acids — Ethyl polyenoate capsule is given as drug intervention. The main components are ethyl eicosapentaenoate (EPA-E) and ethyl docosahexaenoate (DHA-E), both of which will transform into ethyl eicosapentaenoate (EPA) and ethyl docosahexaenoate (DHA). Drug dose is 0.25 g EPA-E&DHA-E; per capsule one at a time, Three times a day.
  Other Names: n-3PUFA
  Arms: n-3PUFA treatment group

SUMMARY:
Crohn's disease (CD) is a chronic recurrent intestinal inflammation involving the whole digestive tract, with high disability rate, high surgical rate and high recurrent rate postoperatively. Preventing postoperative recurrence in CD patients is an important clinical problem needed urgent intervention. Azathioprine (AZA) and infliximab (IFX) effectively prevent postoperative recurrence in CD patients, but the postoperative recurrence rate is still as high as 41%. Oral supplement of n-3 polyunsaturated fatty acids (n-3 PUFA) owns the advantages of high compliance and low economic cost. We aim to evaluate the effect of routine treatment (AZA/IFX) combined with long-term dietary n-3PUFA on the prevention and treatment of postoperative recurrence of CD, which help optimize the treatment strategy for the prevention of postoperative recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. CD patients undergoing partial resection，anastomosis or enterostomy.
2. age ≥18 to ≤80 years;
3. have indications of AZA or IFX application (according to the consensus of ECCO 2016 years);
4. Preoperative diagnosis CD, must provide the biopsy pathological record which accords with the CD diagnosis;
5. If the subject is a woman of childbearing age, pregnancy tests must be conducted at baseline to exclude pregnancy, and the trial process must follow the contraceptive advice of this project
6. subjects must be able and willing to provide written informed consent and comply with the requirements of this research program

Exclusion Criteria:

1. patients without indications use of AZA or IFX;
2. isolated colon CD patients;
3. patients who can't take long-term oral intervention of n-3PUFA;
4. patients diagnosed with short bowel or short bowel syndrome;
5. patients with severe, progressive or uncontrolled kidney, liver, blood or endocrine diseases;
6. postoperative abdominal infection, anastomotic fistula and other complications;
7. there's an infection, Such as Clostridium difficile toxin or other intestinal pathogens infection, active tuberculosis or intestinal tuberculosis, human immunodeficiency virus (HIV) infection, active hepatitis B or hepatitis C;
8. patients with a history of gastrointestinal dysplasia; patients with
9. TPMT gene mutations or low activity;
10. patients who has already participated in other clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2021-02-13 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year postoperative anastomotic recurrence rate | 1 year
  anastomotic recurrence including endoscopic recurrence and imaging recurrence

SECONDARY OUTCOMES:
3 months postoperative anastomotic recurrence rate | 3 months
  anastomotic recurrence including endoscopic recurrence and imaging recurrence
clinical recurrence rate | 3 months，1 year
  CDAI score larger than 150
Inflammatory load | 3 months，1 year
  level of serum C- reactive protein
Inflammatory load | 3 months，1 year
  level of serum fecal calprotectin
Life quality SF-36 | 3 months，1 year
  inflammatory bowel disease questionnaire and health survey summary table SF-36